CLINICAL TRIAL: NCT01546116
Title: Efficacy of Adefovir and Lamivudine Combination Therapy in Patients With Entecavir Resistance
Brief Title: Adefovir and Lamivudine for Entecavir Resistance (ALTER Study)
Acronym: ALTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Hyung Joon Yim, Associate Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER_114093
Record Dates: First submitted 2011-12-22; First posted 2012-03-07 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Hepatitis B
Keywords: adefovir; lamivudine; entecavir resistance
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adefovir and lamivudine combination (Experimental)
  Interventions: Drug: ADEFOVIR, LAMIVUDINE

INTERVENTIONS:
Drug: ADEFOVIR, LAMIVUDINE — Adefovir/10mg tablet/once a day/52week Lamivudine/100mg tablet/once a day/52week
  Other Names: Adefovir (Hepasera); Lamivudine (Zeffix)

SUMMARY:
* Entecavir has been one of the option for treatment of lamivudine resistant chronic hepatitis B (CHB).
* In case of entecavir resistance, adefovir could be used. However, sequential monotherapy may result in multidrug resistance.
* It is thought that adefovir and lamivudine combination therapy reduce the risk of adefovir resistance, thereby continued therapy will lead to suppression of hepatitis B virus (HBV) DNA to be undetectable in patients with entecavir resistance.
* This study aim to evaluate the efficacy of adefovir and lamivudine combination therapy in CHB patients with entecavir resistance.

DETAILED DESCRIPTION:
Entecavir is a potent antiviral agent for the treatment of chronic hepatitis B (CHB). However, the incidence of entecavir resistance increases over 50% at 5th year in lamivudine-refractory CHB patients. Considering cross resistance profile, adefovir is a good option for managing entecavir resistance. However adefovir monotherapy may lead to adefovir resistance, because entecavir resistant hepatitis B virus (HBV) retain lamivudine resistance. Previously, combination of adefovir and lamivudine was reported to be effective in a patient with entecavir resistance, but only as a case report form. No further data are available on this combination therapy in a sufficient number of patients. It is thought that adefovir and lamivudine combination therapy reduce the risk of adefovir resistance, thereby continued combination treatment will result in suppression of HBV DNA to be undetectable in patients with entecavir resistance.

The aim of this study is to evaluate the efficacy of adefovir and lamivudine combination therapy in CHB patients with entecavir resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis B patients (positive HBsAg > 6 months)
2. Age > 18 year old
3. History of treatment with entecavir more than 6 months
4. Proven entecavir resistant mutation (rtT184S/A/I/L/G/C/M, rtS202G/C/I, or rtM250I/V)
5. HBV DNA level> 2000 IU/mL
6. Compensated liver disease (Child-Pugh-Turcotte score over 7; prothrombin time prolonged more than 3 sec above ULN or INR over 1.5; serum albumin >3 g/dL; total bilirubin <2.5 mg/dL; No history of variceal bleeding, ascites, or hepatic encephalopathy)
7. Patients willing to give informed consent

Exclusion Criteria:

1. Out of inclusion criteria
2. Any one of following

   * Serum phosphorus level under 2.4 mg/dL
   * Serum creatinine level over 1.5 mg/dL or creatinine clearance <50 mL/min
   * Absolute neutrophil count lower than 1000 cell/mL
   * Hb level under 10 g/dL (male), under 9 g/dL (female)
   * Serum AFP >100 ng/mL
3. History of treatment with interferon-alfa, thymosin-alfa 1, or nucleos(t)ide analogue other than entecavir in 6 months of screening
4. History of adefovir resistance (detection of rtA181T/Vor rtN236T at screening or in the past)
5. Recipient of organ transplantation
6. Positive antibody test to HIV, HCV or HDV
7. Pregnant or breast feeding women
8. Patients with hepatocellular carcinoma or uncontrolled malignant disease
9. Habitual alcohol drinker (>140 g/week for men, >70 g/week for women) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Degree of HBV DNA reduction from baseline | at week 52
  Degree of HBV DNA reduction from baseline during 52 week-period of adefovir and lamivudine combination therapy will be assessed.

SECONDARY OUTCOMES:
HBV DNA undetectability by PCR (<60 IU/mL) | at week 52
ALT normalization | at week 52
HBeAg loss | at week 52
HBeAg to anti- HBe seroconversion | at week 52
Development of adefovir resistance | at week 52
Virologic breakthrough | at week 52
  virologic breakthrough is defined by increase of HBV DNA above 10 times the lowest level (na dir).

CONTACTS AND LOCATIONS:
Overall Officials: HYUNG JOON YIM, M.D., Ph.D., Principal Investigator — Korea University Ansan Hospital
Locations (9):
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si, Chngcheongbuk-do
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Hallym University, Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - The Catholic University of Korea, Euijeongbu Saint Mary's Hospital, Euijeongbu, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Hallym University, Gangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul

REFERENCES:
- [Background] Lee WM. Hepatitis B virus infection. N Engl J Med. 1997 Dec 11;337(24):1733-45. doi: 10.1056/NEJM199712113372406. No abstract available. PMID 9392700
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Background] Tenney DJ, Rose RE, Baldick CJ, Pokornowski KA, Eggers BJ, Fang J, Wichroski MJ, Xu D, Yang J, Wilber RB, Colonno RJ. Long-term monitoring shows hepatitis B virus resistance to entecavir in nucleoside-naive patients is rare through 5 years of therapy. Hepatology. 2009 May;49(5):1503-14. doi: 10.1002/hep.22841. PMID 19280622
- [Background] Yim HJ, Hussain M, Liu Y, Wong SN, Fung SK, Lok AS. Evolution of multi-drug resistant hepatitis B virus during sequential therapy. Hepatology. 2006 Sep;44(3):703-12. doi: 10.1002/hep.21290. PMID 16941700
- [Background] Lampertico P, Vigano M, Manenti E, Iavarone M, Sablon E, Colombo M. Low resistance to adefovir combined with lamivudine: a 3-year study of 145 lamivudine-resistant hepatitis B patients. Gastroenterology. 2007 Nov;133(5):1445-51. doi: 10.1053/j.gastro.2007.08.079. Epub 2007 Sep 2. PMID 17983801
- [Background] Rapti I, Dimou E, Mitsoula P, Hadziyannis SJ. Adding-on versus switching-to adefovir therapy in lamivudine-resistant HBeAg-negative chronic hepatitis B. Hepatology. 2007 Feb;45(2):307-13. doi: 10.1002/hep.21534. PMID 17256746
- [Result] Villet S, Ollivet A, Pichoud C, Barraud L, Villeneuve JP, Trepo C, Zoulim F. Stepwise process for the development of entecavir resistance in a chronic hepatitis B virus infected patient. J Hepatol. 2007 Mar;46(3):531-8. doi: 10.1016/j.jhep.2006.11.016. Epub 2006 Dec 18. PMID 17239478
- [Result] Yatsuji H, Hiraga N, Mori N, Hatakeyama T, Tsuge M, Imamura M, Takahashi S, Fujimoto Y, Ochi H, Abe H, Maekawa T, Suzuki F, Kumada H, Chayama K. Successful treatment of an entecavir-resistant hepatitis B virus variant. J Med Virol. 2007 Dec;79(12):1811-7. doi: 10.1002/jmv.20981. PMID 17935165